CLINICAL TRIAL: NCT00361777
Title: The Diagnostic Performance of Screening Tests for the Diagnosis of Cushing's Syndrome
Brief Title: Diagnostic Performance of Screening Tests for Cushing s Syndrome
Status: Completed | Type: Observational
Sponsor: Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 020309; 02-CH-0309
Record Dates: First submitted 2006-08-08; First posted 2006-08-09 (Estimated); Last update posted 2019-12-16 (Actual); Status verified 2019-10-30

CONDITIONS: Cushing's Syndrome
Keywords: Dexamethasone; Cushing Syndrome
MeSH Terms: conditions — Cushing Syndrome

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

GROUPS / COHORTS (1):
- Possible Cushing's: Patients with possible cushion's syndrome

SUMMARY:
This study will test the accuracy of screening tests for Cushing s syndrome in overweight people with signs of the disorder. Cushing s syndrome is a rare disorder caused by excess production of the hormone cortisol. Patients may have various problems, such as weight gain, high blood pressure, diabetes, infections, mood problems, trouble concentrating, and increased blood clotting. These symptoms are seen in many other disorders as well, complicating the diagnosis. The reliability of tests currently used to diagnose Cushing s syndrome is not known. To test their accuracy, subjects in this study who test positive for Cushing s syndrome will be evaluated at NIH for 2 years to either confirm or refute the laboratory results.

Patients between 18 and 75 years of age who are being treated at the George Washington University Weight Management Program (GWUWMP) may participate in this study. Candidates will be screened with a medical history, physical examination, measurement of body fat, blood tests, and oral glucose tolerance test. They will also complete a symptoms checklist and quality of life questionnaire.

Participants will be tested for Cushing s syndrome with a saliva collection, 24-hour urine collection, and dexamethasone suppression test (DST). For the DST they will take 1 mg of dexamethasone at night and report to GWUWMP the next morning for a blood draw. All specimens blood, saliva, and urine will be tested for cortisol levels.

People whose test results are abnormal will be seen at the NIH outpatient clinic for a medical history, physical examination, and blood tests; bedtime saliva collection; two 24-hour urine collections; and a 2-day 2-mg DST, followed by administration of corticotropin-releasing hormone (CRH). CRH is a naturally occurring hormone that causes cortisol levels to rise. Pre-treatment with dexamethasone prevents CRH from causing an increase in cortisol in healthy people, but not in patients with Cushing s syndrome. For the 2-day DST, the subject takes 0.5 mg dexamethasone every 6 hours for eight doses. Two hours after the last dose, CRH is injected through a catheter (thin plastic tube) inserted into an arm vein. Blood is drawn just before giving CRH to measure dexamethasone and cortisol levels and after giving CRH to measure cortisol levels.

People whose test results are normal will not be seen further at NIH. Those with high cortisol levels will have repeat urine and saliva tests every 2 to 8 weeks for up to 24 months, and a 1-mg DST every 3 months during routine clinic visits at GWUWMP. People whose increased cortisol is found to be due to another condition besides Cushing s syndrome will be referred for evaluation and possible treatment. Those diagnosed with Cushing s syndrome will have standard tests to identify the tumor causing the disorder, followed by standard medical and surgical treatment.

DETAILED DESCRIPTION:
Cushing's syndrome is a rare disorder characterized by a variety of clinical signs and symptoms that reflect chronic exposure to hypercortisolism such as obesity, hypertension, glucose intolerance, infections, psychiatric disturbance, impaired cognition and hypercoagulability. Thus, it is important to screen for this treatable disorder so as to prevent its associated morbidity and mortality. Because many of the signs of Cushing's syndrome are common in the general population, information about the cost-effectiveness and diagnostic efficiency of various screening tests would be useful.

This study will evaluate the diagnostic performance of various screening tests for Cushing's syndrome in overweight patients recruited from a weight loss center who have additional signs of the disorder. Patients with abnormal tests will be seen as outpatients at the NIH for further evaluation for up to two years to confirm or refute the possibility that they have Cushing's syndrome. Patients with the disorder will be treated.

ELIGIBILITY:
* INCLUSION CRITERIA:

Patients presenting for weight loss treatment at the GWUWMP

Patients must have at least two of the signs and symptoms in Table 1 of the protocol, in addition to weight gain. If abdominal pain, backache and/or headache are present, only one of these symptoms can be used in any given patient, so that another feature must be present.

Willing and able to be seen for up to 24 months

Age 18-75

EXCLUSION CRITERIA:

Weight more than 350 pounds, the maximum weight for radiologist examination tables necessary for the evaluation of Cushing's Syndrome

Renal failure, creatinine greater than 2.6, because of possible effects on dexamethasone metabolism

Pregnancy, because it alters interpretation of adrenal function tests

Current use of oral, inhaled or intranasal glucocorticoids or use within 30 days of study

Other significant medical disorders that may complicate participation or interpretation of the results. For example, a patient with a collagen vascular disorder who has taken intermittent high dose glucocorticoids, and might need to do this again, might not be offered participation.

Use of black licorice or chewing tobacco within two weeks of the study or anticipated use during the study

Use of phenytoin, barbiturate, loperamide or opiates within two weeks of the study or anticipated chronic use during the study.

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 471 (Actual)
Dates: Start 2002-09-19; Study Completion 2019-10-30

PRIMARY OUTCOMES:
Sensitivity and specificity of screening tests | months
  Sensitivity and specificity of screening tests

CONTACTS AND LOCATIONS:
Overall Officials: Lynnette K Nieman, M.D., Principal Investigator — National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK)
Locations (2):
- United States (2):
  - GW University Medical Center GW Hospital Center, Washington D.C., District of Columbia
  - National Institutes of Health Clinical Center, 9000 Rockville Pike, Bethesda, Maryland

REFERENCES:
- [Background] Castro M, Elias PC, Quidute AR, Halah FP, Moreira AC. Out-patient screening for Cushing's syndrome: the sensitivity of the combination of circadian rhythm and overnight dexamethasone suppression salivary cortisol tests. J Clin Endocrinol Metab. 1999 Mar;84(3):878-82. doi: 10.1210/jcem.84.3.5521. PMID 10084565
- [Background] Crapo L. Cushing's syndrome: a review of diagnostic tests. Metabolism. 1979 Sep;28(9):955-77. doi: 10.1016/0026-0495(79)90097-0. PMID 225638
- [Background] Gold PW, Loriaux DL, Roy A, Kling MA, Calabrese JR, Kellner CH, Nieman LK, Post RM, Pickar D, Gallucci W, et al. Responses to corticotropin-releasing hormone in the hypercortisolism of depression and Cushing's disease. Pathophysiologic and diagnostic implications. N Engl J Med. 1986 May 22;314(21):1329-35. doi: 10.1056/NEJM198605223142101. PMID 3010108